CLINICAL TRIAL: NCT04153929
Title: A Phase II, Randomized, Parallel Group, Dose-finding Study of Subcutaneously Administered BI 456906 for 16 Weeks, Compared With Placebo and Open-label Semaglutide in Patients With Type 2 Diabetes Mellitus.
Brief Title: A Study to Test Whether Different Doses of BI 456906 Are Effective in Treating Adults With Type 2 Diabetes.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0002; 2019-002390-60 (EudraCT Number)
Record Dates: First submitted 2019-11-05; First posted 2019-11-06 (Actual); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — BI 456906; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial has a double blind design within each dose group. Patients, investigators and everyone involved in trial conduct or analysis or with any other interest in this trial will remain blinded with regard to the randomized treatment assignments until after database lock. The semaglutide group is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- BI 456906 0.3 mg (Experimental)
  Interventions: Drug: BI 456906
- BI 456906 0.9 mg (Experimental)
  Interventions: Drug: BI 456906
- BI 456906 1.8 mg (Experimental)
  Interventions: Drug: BI 456906
- BI 456906 2.7 mg (Experimental)
  Interventions: Drug: BI 456906
- BI 456906 1.2 twice weekly (2.4) mg (Experimental)
  Interventions: Drug: BI 456906
- BI 456906 1.8 twice weekly (3.6) mg (Experimental)
  Interventions: Drug: BI 456906
- Semaglutide (Active Comparator)
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 456906 — Solution for Injection
  Arms: BI 456906 0.3 mg; BI 456906 0.9 mg; BI 456906 1.2 twice weekly (2.4) mg; BI 456906 1.8 mg; BI 456906 1.8 twice weekly (3.6) mg; BI 456906 2.7 mg
Drug: Placebo — Solution for Injection
  Arms: Placebo
Drug: Semaglutide — Solution for Injection
  Arms: Semaglutide

SUMMARY:
This study is open to adults with type 2 diabetes who take metformin but still have too high blood sugar. The purpose of the study is to find the best dose of BI 456906 that reduces blood sugar. The study also looks at whether BI 456906 helps the participants lose weight.

Participants are in the study for about 23 weeks. During this time, most participants visit the study site about 13 times. Some participants visit the study site about 20 times. At the start of the study, the participants are put into 7 groups. The participants in groups 1 to 6 get injections under the skin once or twice every week. Some participants get different doses of BI 456906 and other participants get placebo. Placebo injections look like the BI 456906 injections, but contain no medicine. Participants in group 7 get semaglutide injections every week. Semaglutide is another medicine for adults with type 2 diabetes.

During the study, the doctors regularly take blood samples from the participants and measure their body weight. The changes in blood sugar levels and body weight are compared between the groups. The doctors also check the general health of the participants.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent in accordance with International conference on harmonization - Good clinical practice (ICH GCP) and local legislation.
* Male and female patients 18 years to 75 years (both inclusive) of age on the day of signing informed consent.
* Diagnosis of Type 2 diabetes mellitus (T2DM) at least 6 months prior to informed consent.
* Glycosylated hemoglobin A1c (HbA1c) 7.0%-10.0% (both inclusive) at screening.
* Treatment with a stable dose of metformin ≥ 1000mg/day for at least 3 months prior to screening.
* Body mass index (BMI) 25 kg/m2-50 kg/m2 (both inclusive) at screening.
* Women of childbearing potential must be ready and able to use highly effective methods of birth control.

Exclusion criteria:

* Patients with type 1 diabetes.
* Exposure to semaglutide, or other Glucagon-like-peptide 1 receptor (GLP-1R) agonists (including combination products) within 3 months prior to screening, or any previous exposure to BI 456906.
* Any additional oral anti-hyperglycemic medication beyond metformin within 3 months prior to screening.
* Use of insulin for glycemic control within 12 months prior to screening.
* Resting Heart Rate >100 bpm or blood pressure ≥160/95 mmHg at screening.
* A marked baseline prolongation of QT/QTc (Fridericia) interval or any other clinically significant Electrocardiogram (ECG) finding at screening.
* Body weight change of +/- 5% or more in the past 3 months or on anti-obesity therapies at any time during the 6 months prior to screening.
* Continuous oral pharmacotherapy to treat any clinical condition during the Trial. Following medications are allowed:

  * metformin, anti-hypertensives (any medication known to cause heart block or bradycardia such as beta-blockers, verapamil and diltiazem are excluded unless used to treat heart rate control or hypertension),
  * Hormone replacement therapy including thyroid hormone, lipid lowering, proton pump inhibitors, H2 blockers for Gastric esophageal reflux disease (GERD), analgesics,
  * sleep medications
  * antihistamines
  * selective Alpha receptor blocker for benign prostatic hyperplasia Patients must be on a stable dose for at least 3 months Prior to Screening
* Any suicidal behavior in the past 2 years, any suicidal ideation of type 4 or 5 in the Columbia-suicide severity rating scale (C-SSRS) in the past 3 months at screening.
* Chronic or relevant acute infections.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (80):
- United States (31):
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Indago Research and Health Center, Hialeah, Florida
  - Meridien Research, Lakeland, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Meridien Research, St. Petersburg, Florida
  - In-Quest Medical Research, LLC, Suwanee, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - DuPage Medical Group, Ltd, Lombard, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - ActivMed Practices & Research, Methuen, Massachusetts
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Mercury Street Medical, Butte, Montana
  - Palm Research Center, Las Vegas, Nevada
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Piedmont Healthcare, Statesville, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Javara Research, Sugar Land, Texas
- Australia (6):
  - Boden Institute of Obesity, Nutrition, Exercies and Eating Disorders, Camperdown, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash University, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
- Austria (2):
  - KH Rudolfstiftung, 1. Med. Abt., Wien, Vienna
  - AKH - Medical University of Vienna, Vienna
- Canada (8):
  - Cook Street Medical Clinic, Victoria, British Columbia
  - LMC Clinical Research Inc. (Brampton), Brampton, Ontario
  - LMC Clinical Research Inc. (Thornhill), Concord, Ontario
  - The Wharton Medical Clinic Clinical Trials Inc., Hamilton, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
  - Manna Research (Quebec), Lévis, Quebec
  - Centre Medical Acadie, Montreal, Quebec
  - Manna Research (Montreal), Pointe-Claire, Quebec
- Czechia (2):
  - Edumed s.r.o, Broumov
  - General Faculty Hospital, Prague, Prague
- Germany (3):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - InnoDiab Forschung GmbH, Essen
  - Institut für Diabetesforschung Münster GmbH, Münster
- Hungary (3):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfured, Balatonfüred
  - Bajcsy-Zsilinszky Hospital and Clinic, Budapest
  - University Debrecen Hospital, Debrecen
- New Zealand (4):
  - Optimal Clinical Trials, Auckland
  - P3 Research, Newtown Wellington NZ
  - P3 Research Kapiti, Paraparaumu
  - P3 Research, Tauranga
- Poland (5):
  - In-Vivo Sp. Z o.o., Bydgoszcz
  - Vita Longa Sp. z o.o., Katowice
  - Pratia SA, Skorzewo
  - Clin.Research Centre Clinsante SC Ewa Galczak-Nowak,Torun, Torun
  - NBR Polska, Warsaw
- GCM Medical Group, PSC, San Juan, Puerto Rico
- South Korea (3):
  - The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si
  - Dongguk University Ilsan Hospital, Goyang
  - Kangdong Sacred Heart Hospital, Seoul
- Spain (4):
  - Hospital A Coruña, A Coruña
  - C.A.P. Sardenya, Barcelona
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clínico de Valencia, Valencia
- Taiwan (3):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
- United Kingdom (5):
  - Waterloo Medical Centre, Blackpool
  - Burbage Surgery, Burbage, Hinkley
  - White Horse Medical Practice, Faringdon
  - Clifton Medical Centre, Rotherham, Rotherham
  - Moorgreen Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Bluher M, Rosenstock J, Hoefler J, Manuel R, Hennige AM. Dose-response effects on HbA1c and bodyweight reduction of survodutide, a dual glucagon/GLP-1 receptor agonist, compared with placebo and open-label semaglutide in people with type 2 diabetes: a randomised clinical trial. Diabetologia. 2024 Mar;67(3):470-482. doi: 10.1007/s00125-023-06053-9. Epub 2023 Dec 14. PMID 38095657
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, multicenter placebo and active comparator controlled, double-blind within dose groups, parallel-group, 16-week trial in patients with type 2 diabetes mellitus (T2DM). An open-label arm (semaglutide) was included as benchmark to compare response curves and support assumptions for Phase III design.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: This arm comprises all placebo treated patients, regardless of the dose group in which they were treated. Patients with type 2 diabetes mellitus with insufficient glycaemic control despite diet, exercise and metformin treatment were administered solution for subcutaneous injection of placebo matched to BI 456906 once weekly for 16 weeks or twice weekly for 16 weeks.
- BI 456906 0.3 mg: Patients with type 2 diabetes mellitus with insufficient glycaemic control despite diet, exercise and metformin treatment were administered once weekly subcutaneously a solution for injection of BI 456906 of 0.3 milligram (mg) on Week 1-Week 16.
- BI 456906 0.9 mg: Patients with type 2 diabetes mellitus with insufficient glycaemic control despite diet, exercise and metformin treatment were administered once weekly subcutaneously a solution for injection of BI 456906 of 0.3 milligram (mg) on Week 1 and Week 2, 0.6 mg on Week 3 and Week 4, 0.9 mg on Week 5-Week 16.
- BI 456906 1.8 mg: Patients with type 2 diabetes mellitus with insufficient glycaemic control despite diet, exercise and metformin treatment were administered once weekly subcutaneously a solution for injection of BI 456906 of 0.3 milligram (mg) on Week 1, 0.6 mg on Week 2, 0.9 mg on Week 3, 1.2 mg on Week 4, 1.5 mg on Week 5, and 1.8 mg on Week 6- Week 16.
- BI 456906 2.7 mg: Patients with type 2 diabetes mellitus with insufficient glycaemic control despite diet, exercise and metformin treatment were administered once weekly subcutaneously a solution for injection of BI 456906 of 0.6 milligram (mg) on Week 1 and Week 2, 1.2 mg on Week 3 and Week 4, 1.8 mg on Week 5, 2.4 mg on Week 6, 2.7 mg on Week 7- Week 16.
- BI 456906 1.2 Twice Weekly (2.4) mg: Patients with type 2 diabetes mellitus with insufficient glycaemic control despite diet, exercise and metformin treatment were administered twice weekly subcutaneously a solution for injection of BI 456906 of 0.3 milligram (mg) on Week 1 and Week 2 (total weekly dose=0.6 mg), 0.6 mg on Week 3 and Week 4 (total weekly dose=1.2 mg), 0.9 mg on Week 5 and Week 6 (total weekly dose=1.8 mg), 1.2 mg on Week 7- Week 16 (total weekly dose 2.4 mg).
- BI 456906 1.8 Twice Weekly (3.6) mg: Patients with type 2 diabetes mellitus with insufficient glycaemic control despite diet, exercise and metformin treatment were administered twice weekly subcutaneously a solution for injection of BI 456906 of 0.3 milligram (mg) on Week 1 (total weekly dose=0.6 mg), 0.6 mg on Week 2 (total weekly dose=1.2 mg), 0.9 mg on Week 3 (total weekly dose=1.8 mg), 1.2 mg on Week 4 (total weekly dose 2.4 mg), 1.5 mg on Week 5 and on Week 6 (total weekly dose 3 mg), 1.8 mg on Week 7 -Week 16 (total weekly dose =3.6 mg).
- Semaglutide: Patients with type 2 diabetes mellitus with insufficient glycaemic control despite diet, exercise and metformin treatment were administered once weekly subcutaneously a solution for injection of Semaglutide of 0.25 milligram (mg) on Week 1-Week 4, 0.5 mg on Week 5-Week 8, 1.0 mg on Week 9-Week 16.
Period: Overall Study
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide
Started (Entered/Randomized) | 60 | 50 | 50 | 52 | 50 | 51 | 50 | 50
Treated | 59 | 50 | 50 | 52 | 50 | 51 | 49 | 50
Completed (Completed planned treatment) | 49 | 41 | 45 | 36 | 33 | 45 | 37 | 45
Not Completed | 11 | 9 | 5 | 16 | 17 | 6 | 13 | 5
Not completed — Other than listed | 2 | 2 | 0 | 1 | 0 | 2 | 2 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 3 | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Adverse Event | 3 | 5 | 5 | 11 | 15 | 4 | 8 | 2
Not completed — Not treated | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS included all patients who were randomized and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide | Total
Number analyzed (Participants) | 59 | 50 | 50 | 52 | 50 | 51 | 49 | 50 | 411
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (10.5) | 56.1 (10.2) | 58.2 (9.6) | 55.3 (10.3) | 59.6 (8.5) | 58.3 (8.8) | 57.7 (9.4) | 55.8 (10.5) | 57.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 22 | 25 | 17 | 24 | 22 | 16 | 178
  Male | 31 | 26 | 28 | 27 | 33 | 27 | 27 | 34 | 233
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 8 | 12 | 12 | 10 | 9 | 14 | 91
  Not Hispanic or Latino | 44 | 39 | 42 | 40 | 38 | 41 | 40 | 36 | 320
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Asian | 8 | 4 | 5 | 8 | 4 | 5 | 3 | 5 | 42
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 3 | 3 | 1 | 2 | 2 | 4 | 3 | 2 | 20
  White | 47 | 42 | 44 | 42 | 43 | 41 | 42 | 43 | 344
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Glycosylated hemoglobin A1c (HbA1c) measured in percentage units [%] [Mean (Standard Deviation); unit: percentage of HbA1c] — Glycosylated hemoglobin A1c (HbA1c) measured in percentage units [%] at baseline is presented.
  percentage of HbA1c | 8.15 (0.85) | 8.09 (0.76) | 7.89 (0.80) | 8.14 (0.86) | 8.18 (0.97) | 8.11 (0.94) | 7.97 (0.71) | 8.03 (0.82) | 8.07 (0.84)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in HbA1c From Baseline to 16 Weeks
Description: Absolute change in glycosylated hemoglobin A1c (HbA1c) from baseline to 16 weeks after treatment start is presented. The measurements for this outcome were performed at baseline and at Week 17.
  Absolute change from baseline in HbA1c to 16 weeks after treatment start was calculated by subtracting the baseline HbA1c value from the HbA1c value at Week 17.
Time Frame: At baseline and at Week 17 (16 weeks after treatment start).
Population: Full Analysis Set (FAS): This patient set included all patients who were randomized and received at least one dose of study drug and who had analysable data for at least one efficacy endpoint. Only patients with non-missing results are reported.
Measure: Mean (Standard Deviation); unit: percentage (%) of HbA1c
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide
Number analyzed (Participants) | 49 | 41 | 46 | 36 | 33 | 44 | 36 | 45
percentage (%) of HbA1c | -0.23 (0.81) | -0.91 (0.71) | -1.37 (0.93) | -1.79 (0.92) | -1.67 (0.78) | -1.68 (0.90) | -1.79 (0.76) | -1.50 (0.84)
Statistical Analysis 1: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; A flat vs. non-flat dose-response relationship across the 6 doses of BI 456906 and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 5 different plausible dose-response patterns (linear, exponential, Emax 1, Emax 2 and Sigmoid Emax) while protecting the overall probability of type I error (one-sided alpha of 0.025). For the twice weekly dosing schemes the total dose per week was considered for the MCP-Mod analysis; Test type: Other — Mixed Model Repeated Measures (MMRM) estimates were used as input for the MCP-Mod. MMRM with fixed, categorical factors of treatment at each visit, and continuous factors of baseline at each visit, using visit (Week 5, 8, 12, 16 and 17) as repeated measures, subject as random effect, unstructured covariance matrix to model within subject measurements; p < 0.0001, MCP-Mod linear model fit; Model assumption: The maximum effect is achieved at 3.6 mg dose
Statistical Analysis 2: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, MCP-Mod Exponential model fit; Model assumption: 90% of the maximum effect is achieved at 3.6 mg dose
Statistical Analysis 3: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, MCP-Mod Emax 1 model fit; Model assumption: 90% of the maximum effect is achieved at 3.6 mg dose
Statistical Analysis 4: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, MCP-Mod Emax 2 model fit; Model assumption: 70% of the maximum effect is achieved at 3.6 mg dose
Statistical Analysis 5: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, MCP-Mod Sigmoid Emax model fit; Model assumption: 50% of the maximum effect is achieved at 1.8 mg and 90% of the maximum effect is achieved at 3.6 mg dose
Statistical Analysis 6: Comparison: Placebo vs BI 456906 0.3 mg; Mixed Model Repeated Measures (MMRM) with fixed, categorical factors of treatment at each visit, and continuous factors of baseline at each visit, using visit (Week 5, 8, 12, 16 and 17) as repeated measures, subject as random effect, unstructured covariance matrix to model within subject measurements; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -0.76, 95% CI 2-sided [-1.06 to -0.46] — Difference was calculated as BI 456906 0.3 mg - Placebo at Week 17
Statistical Analysis 7: Comparison: Placebo vs BI 456906 0.9 mg; [analysis description as in outcome 1, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -1.31, 95% CI 2-sided [-1.60 to -1.01] — Difference was calculated as BI 456906 0.9 mg - Placebo at Week 17
Statistical Analysis 8: Comparison: Placebo vs BI 456906 1.8 mg; [analysis description as in outcome 1, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -1.56, 95% CI 2-sided [-1.87 to -1.26] — Difference was calculated as BI 456906 1.8 mg - Placebo at Week 17
Statistical Analysis 9: Comparison: Placebo vs BI 456906 2.7 mg; [analysis description as in outcome 1, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -1.41, 95% CI 2-sided [-1.72 to -1.10] — Difference was calculated as BI 456906 2.7 mg - Placebo at Week 17
Statistical Analysis 10: Comparison: Placebo vs BI 456906 1.2 Twice Weekly (2.4) mg; [analysis description as in outcome 1, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -1.49, 95% CI 2-sided [-1.78 to -1.19] — Difference was calculated as "BI 456906 1.2 twice weekly (2.4) mg" - "Placebo" at Week 17
Statistical Analysis 11: Comparison: Placebo vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -1.53, 95% CI 2-sided [-1.84 to -1.22] — Difference was calculated as "BI 456906 1.8 twice weekly (3.6) mg" - "Placebo" at Week 17

2. Secondary Outcome: Key Secondary Endpoint: The Relative Change in Body Weight From Baseline to 16 Weeks
Description: The relative change in body weight from baseline to 16 weeks after treatment start is presented. The measurements for this outcome were performed at baseline and at Week 17.
  The relative change in body weight from baseline to 16 weeks after treatment start was calculated as (body weight at Week 17 - body weight at baseline/body weight at baseline) * 100.
Time Frame: At baseline and at Week 17 (16 weeks after treatment start ).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body weight change
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide
Number analyzed (Participants) | 49 | 41 | 46 | 36 | 33 | 44 | 37 | 45
percentage of body weight change | -1.20 (3.52) | -1.86 (2.91) | -4.43 (3.92) | -6.63 (5.13) | -6.68 (4.05) | -7.16 (6.06) | -8.95 (5.33) | -5.40 (4.33)
Statistical Analysis 1: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — Mixed Model Repeated Measures (MMRM) estimates were used as input for the MCP-Mod. MMRM with fixed, categorical factors of treatment at each visit, and continuous factors of baseline at each visit, using visit (Week 2, 3, 4, 5, 6, 7, 8, 12, 16 and 17 ) as repeated measures, subject as random effect, unstructured covariance matrix to model within subject measurements; p < 0.0001, MCP-Mod linear model fit; Model assumption: The maximum effect is achieved at 3.6 mg dose
Statistical Analysis 2: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, MCP-Mod exponential model fit; Model assumption: 90% of the maximum effect is achieved at 3.6 mg dose
Statistical Analysis 3: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, MCP-Mod Emax 1 model fit; Model assumption: 90% of the maximum effect is achieved at 3.6 mg dose
Statistical Analysis 4: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, MCP-Mod Emax 2 model fit; Model assumption: 70% of the maximum effect is achieved at 3.6 mg dose
Statistical Analysis 5: Comparison: Placebo vs BI 456906 0.3 mg vs BI 456906 0.9 mg vs BI 456906 1.8 mg vs BI 456906 2.7 mg vs BI 456906 1.2 Twice Weekly (2.4) mg vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, MCP-Mod Sigmoid Emax model fit; [statistical method as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Placebo vs BI 456906 0.3 mg; Mixed Model Repeated Measures (MMRM) with fixed, categorical factors of treatment at each visit, and continuous factors of baseline at each visit, using visit (Week 2, 3, 4, 5, 6, 7, 8, 12, 16 and 17 ) as repeated measures, subject as random effect, unstructured covariance matrix to model within subject measurements; Test type: Other — No formal hypotheses were tested; p = 0.2228, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -1.11, 95% CI 2-sided [-2.90 to 0.68] — Difference was calculated as "BI 456906 0.3 mg" - "Placebo" at Week 17
Statistical Analysis 7: Comparison: Placebo vs BI 456906 0.9 mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -3.79, 95% CI 2-sided [-5.56 to -2.01] — Difference was calculated as "BI 456906 0.9 mg" - "Placebo" at Week 17
Statistical Analysis 8: Comparison: Placebo vs BI 456906 1.8 mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -5.61, 95% CI 2-sided [-7.41 to -3.81] — Difference was calculated as "BI 456906 1.8 mg" - "Placebo" at Week 17
Statistical Analysis 9: Comparison: Placebo vs BI 456906 2.7 mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -6.25, 95% CI 2-sided [-8.12 to -4.38] — Difference was calculated as "BI 456906 2.7 mg" - "Placebo" at Week 17
Statistical Analysis 10: Comparison: Placebo vs BI 456906 1.2 Twice Weekly (2.4) mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -6.25, 95% CI 2-sided [-8.02 to -4.47] — Difference was calculated as "BI 456906 1.2 twice weekly (2.4) mg" - "Placebo" at Week 17
Statistical Analysis 11: Comparison: Placebo vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -7.68, 95% CI 2-sided [-9.52 to -5.83] — Difference was calculated as "BI 456906 1.8 twice weekly (3.6) mg" - "Placebo" at Week 17

3. Secondary Outcome: The Absolute Change in Body Weight From Baseline to 16 Weeks
Description: The absolute change in body weight from baseline to 16 weeks after treatment start is presented. Measurements for this outcome were performed at baseline and at Week 17.
  The absolute change in body weight from baseline to 16 weeks after treatment start was calculated as: body weight at Week 17- body weight at baseline.
Time Frame: At baseline and at Week 17 (16 weeks after treatment start).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide
Number analyzed (Participants) | 49 | 41 | 46 | 36 | 33 | 44 | 37 | 45
kilogram (kg) | -1.28 (3.05) | -1.90 (3.12) | -4.41 (4.07) | -6.31 (4.53) | -6.88 (4.41) | -6.75 (6.10) | -8.88 (4.93) | -5.18 (4.52)
Statistical Analysis 1: Comparison: Placebo vs BI 456906 0.3 mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p = 0.4439, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -0.66, 95% CI 2-sided [-2.34 to 1.03] — Difference was calculated as "BI 456906 0.3 mg" - "Placebo" at Week 17
Statistical Analysis 2: Comparison: Placebo vs BI 456906 0.9 mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p = 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -3.28, 95% CI 2-sided [-4.95 to -1.61] — Difference was calculated as "BI 456906 0.9 mg" - "Placebo" at Week 17
Statistical Analysis 3: Comparison: Placebo vs BI 456906 1.8 mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -4.93, 95% CI 2-sided [-6.62 to -3.23] — Difference was calculated as "BI 456906 1.8 mg" - "Placebo" at Week 17
Statistical Analysis 4: Comparison: Placebo vs BI 456906 2.7 mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -5.76, 95% CI 2-sided [-7.53 to -4.00] — Difference was calculated as "BI 456906 2.7 mg" - "Placebo" at Week 17
Statistical Analysis 5: Comparison: Placebo vs BI 456906 1.2 Twice Weekly (2.4) mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -5.44, 95% CI 2-sided [-7.11 to -3.77] — Difference was calculated as "BI 456906 1.2 twice weekly (2.4) mg" - "Placebo" at Week 17
Statistical Analysis 6: Comparison: Placebo vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -7.05, 95% CI 2-sided [-8.79 to -5.31] — Difference was calculated as "BI 456906 1.8 twice weekly (3.6) mg" - "Placebo" at Week 17
Statistical Analysis 7: Comparison: Placebo vs Semaglutide; [analysis description as in outcome 2, analysis 6]; Test type: Other — No formal hypotheses were tested; p < 0.0001, Mixed Model Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -3.85, 95% CI 2-sided [-5.52 to -2.18] — Difference was calculated as "Semaglutide" - "Placebo" at Week 17

4. Secondary Outcome: The Absolute Change in Waist Circumference From Baseline to 16 Weeks
Description: The absolute change in waist circumference from baseline to 16 weeks after treatment start is presented. Measurements for this outcome were performed at baseline and at Week 17.
  The absolute change in waist circumference from baseline to 16 weeks after treatment start was calculated as: waist circumference at Week 17- waist circumference at baseline.
Time Frame: At baseline and at Week 17 (16 weeks after treatment start).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide
Number analyzed (Participants) | 49 | 43 | 47 | 39 | 35 | 45 | 36 | 46
centimeter | -1.95 (9.08) | -2.73 (10.49) | -1.80 (10.55) | -3.63 (10.94) | -7.47 (12.24) | -4.61 (9.73) | -12.89 (25.50) | -3.63 (5.05)
Statistical Analysis 1: Comparison: Placebo vs BI 456906 0.3 mg; Mixed Model Repeated Measures (MMRM) with fixed, categorical factors of treatment at each visit, and continuous factors of baseline at each visit, using visit (Week 6 and 17 ) as repeated measures, subject as random effect, unstructured covariance matrix to model within subject measurements; Test type: Other — No formal hypotheses were tested; p = 0.7708, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -0.62, 95% CI 2-sided [-4.82 to 3.57] — Difference was calculated as "BI 456906 0.3 mg" - "Placebo" at Week 17
Statistical Analysis 2: Comparison: Placebo vs BI 456906 0.9 mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.7462, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = 0.68, 95% CI 2-sided [-3.44 to 4.79] — Difference was calculated as "BI 456906 0.9 mg" - "Placebo" at Week 17
Statistical Analysis 3: Comparison: Placebo vs BI 456906 1.8 mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.1302, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -3.32, 95% CI 2-sided [-7.62 to 0.98] — Difference was calculated as "BI 456906 1.8 mg" - "Placebo" at Week 17
Statistical Analysis 4: Comparison: Placebo vs BI 456906 2.7 mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.0414, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -4.61, 95% CI 2-sided [-9.03 to -0.18] — Difference was calculated as "BI 456906 2.7 mg" - "Placebo" at Week 17
Statistical Analysis 5: Comparison: Placebo vs BI 456906 1.2 Twice Weekly (2.4) mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.2273, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -2.55, 95% CI 2-sided [-6.71 to 1.60] — Difference was calculated as "BI 456906 1.2 twice weekly (2.4) mg" - "Placebo" at Week 17
Statistical Analysis 6: Comparison: Placebo vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.0002, Mixed Model for Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -8.40, 95% CI 2-sided [-12.81 to -3.98] — Difference was calculated as "BI 456906 1.8 twice weekly (3.6) mg" - "Placebo" at Week 17
Statistical Analysis 7: Comparison: Placebo vs Semaglutide; [analysis description as in outcome 4, analysis 1]; Test type: Other — No formal hypotheses were tested; p = 0.1967, Mixed Model Repeated Measures (MMRM) — P-value is considered nominal; Kenward-Roger was used to estimate denominator degrees of freedom; Difference of adjusted means = -2.72, 95% CI 2-sided [-6.86 to 1.42] — Difference was calculated as "Semaglutide" - "Placebo" at Week 17

5. Secondary Outcome: Percentage of Patients With 5 % or Greater Body Weight Loss From Baseline to 16 Weeks
Description: The percentage of patients with 5 percent (%) or greater body weight loss from baseline to 16 weeks after treatment start is presented.
  Measurements for this outcome were performed at baseline and at Week 17.
Time Frame: At baseline and at Week 17 (16 weeks after treatment start).
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide
Number analyzed (Participants) | 59 | 50 | 50 | 52 | 50 | 51 | 49 | 50
percentage of patients | 6.8 | 8.0 | 38.0 | 42.3 | 46.0 | 56.9 | 57.1 | 38.0
Statistical Analysis 1: Comparison: Placebo vs BI 456906 0.3 mg; Method: Logistic regression model for body weight loss with treatment as fixed effect; Test type: Other; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.28 to 5.20] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 2: Comparison: Placebo vs BI 456906 0.9 mg; Method: Logistic regression model for body weight loss with treatment as fixed effect; Test type: Other; Odds Ratio (OR) = 7.92, 95% CI 2-sided [2.43 to 25.74] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 3: Comparison: Placebo vs BI 456906 1.8 mg; Method: Logistic regression model for body weight loss with treatment as fixed effect; Test type: Other; Odds Ratio (OR) = 17.68, 95% CI 2-sided [5.21 to 60.03] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 4: Comparison: Placebo vs BI 456906 2.7 mg; Method: Logistic regression model for body weight loss with treatment as fixed effect; Test type: Other; Odds Ratio (OR) = 25.87, 95% CI 2-sided [7.31 to 91.55] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 5: Comparison: Placebo vs BI 456906 1.2 Twice Weekly (2.4) mg; Method: Logistic regression model for body weight loss with treatment as fixed effect; Test type: Other; Odds Ratio (OR) = 21.75, 95% CI 2-sided [6.57 to 72.04] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 6: Comparison: Placebo vs BI 456906 1.8 Twice Weekly (3.6) mg; Method: Logistic regression model for body weight loss with treatment as fixed effect; Test type: Other; Odds Ratio (OR) = 35.00, 95% CI 2-sided [9.84 to 124.47] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 7: Comparison: Placebo vs Semaglutide; Method: Logistic regression model for body weight loss with treatment as fixed effect; Test type: Other; Odds Ratio (OR) = 8.22, 95% CI 2-sided [2.52 to 26.79] — Odds Ratio was calculated as Semaglutide / Placebo

6. Secondary Outcome: Percentage of Patients With 10% or Greater Body Weight Loss From Baseline to 16 Weeks
Description: The percentage of patients with 10 % or greater body weight loss from baseline to 16 weeks after treatment start is presented.
  Measurements for this outcome were performed at baseline and at Week 17.
Time Frame: At baseline and at Week 17 (16 weeks after treatment start).
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide
Number analyzed (Participants) | 59 | 50 | 50 | 52 | 50 | 51 | 49 | 50
percentage of patients | 0.0 | 2.0 | 6.0 | 13.5 | 16.0 | 25.5 | 34.7 | 16.0
Statistical Analysis 1: Comparison: Placebo vs BI 456906 0.3 mg; Method: Logistic regression model using Firth's bias-reducing penalized maximum likelihood estimation for body weight loss with treatment as fixed effect; Test type: Other; Odds Ratio (OR) = 3.67, 95% CI 2-sided [0.14 to 95.73] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 2: Comparison: Placebo vs BI 456906 0.9 mg; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 7.97, 95% CI 2-sided [0.39 to 163.56] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 3: Comparison: Placebo vs BI 456906 1.8 mg; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 25.17, 95% CI 2-sided [1.35 to 471.09] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 4: Comparison: Placebo vs BI 456906 2.7 mg; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 33.01, 95% CI 2-sided [1.78 to 613.51]
Statistical Analysis 5: Comparison: Placebo vs BI 456906 1.2 Twice Weekly (2.4) mg; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 42.44, 95% CI 2-sided [2.37 to 761.44] — Odds Ratio was calculated as BI 456906 / Placebo
Statistical Analysis 6: Comparison: Placebo vs BI 456906 1.8 Twice Weekly (3.6) mg; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 84.53, 95% CI 2-sided [4.71 to 999] — Odds Ratio was calculated as BI 456906 / Placebo. The upper limit is bigger than 999
Statistical Analysis 7: Comparison: Placebo vs Semaglutide; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 22.44, 95% CI 2-sided [1.22 to 413.33] — Odds Ratio was calculated as Semaglutide / Placebo

ADVERSE EVENTS:
Time Frame: From first intake of any trial drug until last intake of any trial drug (planned: 16 weeks) + residual effect period (BI 456906: 28 days, Semaglutide: 35 days), up to 159 days.
Description: Treated set (TS): This patient set included all patients who were randomized and received at least one dose of study drug.
Arm/Group | Placebo | BI 456906 0.3 mg | BI 456906 0.9 mg | BI 456906 1.8 mg | BI 456906 2.7 mg | BI 456906 1.2 Twice Weekly (2.4) mg | BI 456906 1.8 Twice Weekly (3.6) mg | Semaglutide
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/50 | 0/50 | 0/52 | 0/50 | 0/51 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/59 | 1/50 | 4/50 | 3/52 | 2/50 | 1/51 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 18/59 | 27/50 | 30/50 | 40/52 | 33/50 | 33/51 | 37/49 | 20/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | BI 456906 0.3 mg (N=50) | BI 456906 0.9 mg (N=50) | BI 456906 1.8 mg (N=52) | BI 456906 2.7 mg (N=50) | BI 456906 1.2 Twice Weekly (2.4) mg (N=51) | BI 456906 1.8 Twice Weekly (3.6) mg (N=49) | Semaglutide (N=50)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune disorder (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | BI 456906 0.3 mg (N=50) | BI 456906 0.9 mg (N=50) | BI 456906 1.8 mg (N=52) | BI 456906 2.7 mg (N=50) | BI 456906 1.2 Twice Weekly (2.4) mg (N=51) | BI 456906 1.8 Twice Weekly (3.6) mg (N=49) | Semaglutide (N=50)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 6 | 2 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 1 | 5 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 2 | 7 | 7 | 8 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 12 | 8 | 9 | 7 | 8 | 11 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 3 | 5 | 4 | 4 | 7 | 1
Eructation (Gastrointestinal disorders) | 0 | 2 | 2 | 3 | 3 | 1 | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 2 | 3 | 2 | 1 | 4 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 3 | 4 | 2 | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 5 | 10 | 14 | 25 | 23 | 14 | 23 | 6
Vomiting (Gastrointestinal disorders) | 3 | 7 | 9 | 12 | 13 | 6 | 11 | 2
Asthenia (General disorders) | 0 | 1 | 2 | 3 | 1 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 3 | 1 | 3 | 2 | 4 | 5 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 2 | 1 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 4 | 2 | 1 | 1 | 1
Lipase increased (Investigations) | 0 | 2 | 4 | 1 | 2 | 1 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 6 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6 | 7 | 6 | 11 | 9 | 15 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 3 | 2 | 0 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3 | 2 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 4 | 0 | 1 | 1 | 3 | 1
Headache (Nervous system disorders) | 4 | 4 | 5 | 4 | 1 | 3 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT04153929/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT04153929/SAP_001.pdf